CLINICAL TRIAL: NCT03276065
Title: Randomized Controlled Trial of Laser Hair Depilation in Adolescents With Pilonidal Disease
Brief Title: Effectiveness of Laser Hair Removal in Pilonidal Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Peter Minneci, Associate Professor of Surgery and Pediatrics, Nationwide Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB17-00186
Record Dates: First submitted 2017-09-05; First posted 2017-09-08 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Pilonidal Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Laser plus Standard of Care Depilation (Experimental): Laser depilation to the natal cleft (pilonidal region) every 4-6 weeks for 5 treatments with either an 810nm or Nd:YAG laser dependent on Fitzpatrick skin type and tolerability. Patients and families in the intervention group will also be taught hair removal techniques and asked to perform either chemical or mechanical depilation as needed to keep the area hair-free between clinic treatments.
  Interventions: Device: Laser depilation
- Standard of Care Depilation (Active Comparator): Patients and families in the standard of care group will be taught hair removal techniques and asked to perform either chemical or mechanical depilation as needed to keep the area hair-free. Patients will be given supplies for six months of hair removal.
  Interventions: Other: Standard of care hair depilation

INTERVENTIONS:
Device: Laser depilation — Fitzpatrick skin type classification will be assessed during the initial visit. The Fitzpatrick skin type classification is based on the level of pigmentation of the skin and its response to ultraviolet light (See Appendix). It will be used to select the best laser to perform hair removal for each patient. The laser treatment group will consist of an 810 nm (for Fitzpatrick skin types I-IV) or Nd:YAG (for Fitzpatrick skin types V-VI) 28 joule application at auto pulse duration for 400 ms. A cooling platform and application of 7% lidocaine/ 7% tetracaine cream, applied 45 minutes prior to treatment, will minimize any discomfort associated with the heat of the laser treatments.
  Arms: Laser plus Standard of Care Depilation
Other: Standard of care hair depilation — Patients and families in the standard of care group will be taught hair removal techniques and asked to perform either chemical or mechanical depilation as needed to keep the area hair-free. Patients will be given supplies for six months of hair removal.
  Arms: Standard of Care Depilation

SUMMARY:
Pilonidal disease is a common painful condition that affects 26 per 100,000 people with an incidence of 1.1% in the young male population. Recurrence rates of pilonidal disease after initial incision and drainage and after resection have been reported to be 16% and 11% respectively. Furthermore, wound issues after resection with primary closure have been reported to be as high as 30%. In several retrospective studies and small prospective studies, laser hair removal has shown promise as an adjunct therapy to decrease recurrent infections and decrease the need for repeat surgery in adults and older adolescents. We are performing a randomized control trial of laser hair depilation plus chemical/mechanical depilation to examine outcomes related to recurrence of pilonidal disease.

ELIGIBILITY:
Inclusion Criteria:

* All Fitzpatrick skin types
* 11-21 years of age
* Diagnosis of pilonidal disease

Exclusion Criteria:

* History of photosensitivity
* Actively inflamed pilonidal sinus. These patients are invited to participate upon resolution of their inflamed sinus.

Ages: 11 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 302 (Estimated)
Dates: Start 2017-09-05 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Recurrence of pilonidal disease | 12 months
  Recurrence is defined as a new development of pilonidal abscess, folliculitis, or draining sinus after treatment which would require antibiotic treatment, additional surgical incision and drainage or excision.

SECONDARY OUTCOMES:
Disability Days | 12 months
  Defined as days that patient does participate in all normal activities due to their pilonidal disease
Health related quality of life | 1 year
  Measured using PedsQL scales

CONTACTS AND LOCATIONS:
Overall Officials: Peter C Minneci, MD, MHSc, Principal Investigator — Nationwide Children's Hospital; Katherine J Deans, MD, MHSc, Study Director — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

REFERENCES:
- [Derived] Minneci PC, Gil LA, Cooper JN, Asti L, Nishimura L, Lutz CM, Deans KJ. Laser Epilation as an Adjunct to Standard Care in Reducing Pilonidal Disease Recurrence in Adolescents and Young Adults: A Randomized Clinical Trial. JAMA Surg. 2024 Jan 1;159(1):19-27. doi: 10.1001/jamasurg.2023.5526. PMID 37938854
- [Derived] Minneci PC, Halleran DR, Lawrence AE, Fischer BA, Cooper JN, Deans KJ. Laser hair depilation for the prevention of disease recurrence in adolescents and young adults with pilonidal disease: study protocol for a randomized controlled trial. Trials. 2018 Nov 1;19(1):599. doi: 10.1186/s13063-018-2987-7. PMID 30382903